CLINICAL TRIAL: NCT07258524
Title: PET Assessment of Disease Activity and Cardiovascular Disease Risk in ANCA-associated Vasculitis
Acronym: PANDA-VASC
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC25078
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: ANCA Associated Vasculitis (AAV)
Keywords: ANCA; Vasculitis; PET scanning
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vasculitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ANCA associated vasculitis (AAV) group: All participants will have a diagnosis of ANCA-associated vasculitis (AAV) in accordance with the 2012 Revised International Chapel Hill Consensus Conference Nomenclature of Vasculitides criteria and clinician's assessment. At enrolment, participants in the AAV group will have active disease, as defined by the presence of symptoms and signs attributable to active vasculitis necessitating the commencement or increase in immunosuppressive treatment other than glucocorticoids.
  In order to return for the follow-up visit, participants will be in clinical remission. Remission will be defined as Birmingham Vasculitis Activity Score (BVAS) = 0 for at least two months whilst taking prednisolone at a daily of dose ≤7.5mg in conjunction with the treating clinician's assessment of clinically silent disease.
- Matched control group: All participants will be matched with the AAV group based on age, gender, ethnicity, and cardiovascular disease risk factors including impaired kidney function. They will have no additional health problems and be taking no additional medications (other than those relevant to cardiovascular disease risk) that may interfere with PET imaging.

SUMMARY:
Antineutrophil cytoplasm antibody (ANCA)-associated vasculitis (AAV) is a severe autoimmune condition characterised by inflammation of small blood vessels. The condition causes multi-organ dysfunction and, if left untreated, is usually fatal. AAV is difficult to diagnose and the degree of disease activity is challenging to monitor. Current methods of disease activity assessment are either inaccurate (blood tests), invasive (biopsy), or non-specific (imaging). Additionally, though modern treatments are effective, patients with AAV remain at a substantially increased risk of cardiovascular disease (CVD) in the long-term. There is therefore an urgent need for a tool which is able to reliably identify disease, and assess long-term CVD risk.

Total-Body PET imaging with FDG, DOTATATE, and FAPI radiotracers may provide the answer. This study will recruit patients with active AAV, together with a control group of individuals without the disease, to undergo Total-Body FDG, DOTATATE, and FAPI PET scanning and compare the results with established measures of disease activity and CVD risk assessment.

The investigators believe that Total-Body PET scanning will be capable of accurately identifying AAV disease and those at increased CVD risk. This could enhance understanding and improve the management of those with the condition.

This study will recruit a group of patients with AAV and a comparator groups of 'matched' individuals without AAV. Comparisons between groups will allow the investigators to ensure that the changes seen are due to AAV disease. The study will recruit a minimum of 30 and a maximum of 90 participants in the AAV group, and a minimum of 10 and maximum of 30 participants in the matched control group.

AAV subjects and matched control subjects will undergo baseline total-body PET scanning with either one, two or three radiotracers ([18F]-FDG, [68Ga]-DOTATATE, and [68Ga]-FAPI). Alongside this they will receive assessment of cardiovascular disease risk including 24-hour blood pressure measurement, arterial stiffness measurement, and retinal scanning. Participants will also supply a blood and urine sample.

For matched control subjects, their participation will end at this point. Subjects in the AAV group will undergo repeat assessment with total-body PET imaging and cardiovascular disease risk measurement once their condition is in remission (usually after around 3-6 months).

The investigators will compare PET scan results between groups, and with cardiovascular assessments. This will allow determination of whether total-body PET scanning can identify AAV disease activity, and whether it can inform CVD risk.

All research activity will be carried out within the University of Edinburgh BioQuarter, including the Royal infirmary of Edinburgh, the Edinburgh Imaging Facility, and Queen's Medical Research Institute.

DETAILED DESCRIPTION:
Antineutrophil cytoplasm antibody (ANCA)-associated vasculitis (AAV) is a rare condition which causes widespread blood vessel inflammation, leading to dysfunction in several organs. The condition is autoimmune, meaning that it is driven by an abnormal response from the body's own immune system, though the exact cause is unknown. Without treatment most patients with AAV will die. However current treatment is effective, with ~90% of patients alive at 1-year following diagnosis. Once the initial phase of the disease is controlled, patients remain at risk of relapse which can be difficult to detect. Additionally, in the long term, patients remain at an increased risk of death as a result of cardiovascular disease (CVD), including heart attacks and strokes.

The diagnosis of AAV is challenging and often delayed, meaning established organ damage is often present at diagnosis. Accurate assessment of disease activity is essential to guide best treatment in AAV. Smouldering, unchecked inflammation contributes to morbidity and to the development of CVD. Conversely, attributing symptoms to active disease when they are due to established injury risks overtreatment and associated side effects, which can be significant.

Current methods of disease activity assessment are limited. Biopsy is considered the gold standard, however, can only assess disease in one organ at a time, and is an invasive and unpleasant test. Several scans are currently available, though each is also limited in terms of coverage and accuracy. Accordingly, new methods of disease activity assessment are required which provide an accurate, non-invasive, and multi-system approach, both at presentation and throughout the disease course.

Additionally, even when disease control is optimum, patients with AAV remain at an increased risk of CVD. Methods to identify those at the highest risk of CVD events are lacking, thus personalising preventative therapies remains a challenge. Tools that can highlight those at an increased risk of CVD events are urgently needed.

Total-Body positron emission tomography (PET) scanning provides a potential solution to both of these problems.

PET scanning allows detection and quantification of disease within the body. With the advent of Total-Body PET facilities, scans now benefit from enhanced coverage, accuracy, and speed. Patients can now be reliably scanned from 'top to toe' relatively quickly, and with an acceptable degree of radiation exposure. Despite being used in several similar conditions, PET has never been adequately assessed in AAV.

PET scanning requires the injection of a 'radiotracer' which binds to areas of disease and can then be picked up by the scanner. Historically, we have used a radiotracer called FDG, however a number of newer radiotracers are now available which may be more accurate. The radiotracer DOTATATE may bind more specifically to the inflammation caused by AAV, allowing a more accurate picture of the disease to be painted. Additionally, the radiotracer FAPI finds to areas of fibrosis, or scarring. this radiotracer therefore has the potential to tell us about a different aspect of the disease, and help differentiate active inflammation from tissue damage and remodelling.

Finally, in addition to identifying active AAV disease, both FDG and DOTATATE may be able to inform which patients are more at risk of developing CVD in the future.

Accordingly, this study aims to assess the ability of Total-Body PET scanning, using three different radiotracers, to accurately assess disease activity in AAV, and identify those patients at an increased risk of CVD in the long term. This would improve outcomes for these patients, and increase understanding of the condition.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years of age
2. Diagnosis of active AAV (AAV group)

Exclusion Criteria:

1. Outwith early treatment window (must receive baseline scan <3 weeks from starting treatment)
2. Pregnancy or breastfeeding
3. Advanced renal dysfunction (eGFR <15ml/min/1.73m2)
4. Adverse reaction or hypersensitivity to proposed radiotracers
5. Insulin-dependent diabetes mellitus
6. Patients without mental capacity or willingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AAV group: all participants will have a diagnosis of ANCA-associated vasculitis (AAV) in accordance with the 2012 Revised International Chapel Hill Consensus Conference Nomenclature of Vasculitides criteria and clinician's assessment. At enrolment, participants in the AAV group will have active disease, as defined by the presence of symptoms and signs attributable to active vasculitis necessitating the commencement or increase in immunosuppressive treatment other than glucocorticoids.
  Matched control group: all participants will be matched with the AAV group based on age, gender, ethnicity, and cardiovascular disease risk factors including impaired kidney function. They will have no additional health problems and be taking no additional medications (other than those relevant to cardiovascular disease risk) that may interfere with PET imaging.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Change in tracer ([18F]-FDG, [68Ga]-DOTATATE, and [68Ga]-FAPI) uptake (calculated using maximum standardised uptake values (SUVmax)) within regions of interest between baseline and remission) | 3-12 months
  The change in PET radiotracer uptake within regions of interest between patients with active AAV (e.g. at baseline) and patients in remission (e.g. at follow-up)

SECONDARY OUTCOMES:
Correlation between tracer uptake (SUVmax and SUVmean) and established measures of disease activity including: o CRP o ANCA titre o Patient reported disease activity o Physician estimated disease activity | 3-12 months
  As above
Correlation between tracer uptake (SUVmax and SUVmean) and established surrogate measures of CVD risk including: o Arterial stiffness o 24-hour ambulatory blood pressure o Retinal OCT imaging metrics | 3-12 months
  As above

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Dhaun, MBChB PhD, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No